CLINICAL TRIAL: NCT02518386
Title: Evaluation of the Epidemiology and the Take Load of Voluntary Drug Intoxications by the Emergency Structures in France
Brief Title: Epidemiology of Acute Self-poisoning in Emergency Services in France
Acronym: EpiTox
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: French Society of Emergency Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: EpiTox
Record Dates: First submitted 2015-02-24; First posted 2015-08-07 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Suicide Attempts
Keywords: emergency department; epidemiology; prehospital care; dispatch; acute self poisoning
MeSH Terms: conditions — Suicide, Attempted; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — No intervention is planned

SUMMARY:
Acute self poisoning is a leading cause of suicide attempts and leads to frequent emergency department visits. However, the exact epidemiology of acute self poisoning is not known. The description of the clinical pathway and the characteristics of patients with acute self poisoning could lead to an improvement in emergency care.

The Investigators will conduct a 48h observational study in emergency services in France. Investigators primary objective is to gathered epidemiological clinical and treatment data during emergency dispatch, prehospital care and inhospital emergency care.

DETAILED DESCRIPTION:
Acute self poisoned patients will be prospectively and anonymously recruited by emergency physicians in charge during two days. Acute self poisoning is define as follow: intentional medicine intake in the 24h hours before emergency department admission.

Epidemiological, clinical, toxicological and treatment data will be gathered. Outcome of patient will be prospectively assessed at 30days.

All data will be transmitted to the principal investigators. Then, 20% of the data will be monitored by an independent committee.

Exhaustivity will be retrospectively assessed by the number of inclusions in 10 emergency centers divided by the total number of possible inclusions in these centers.

Finally, an independent statistician will be in charge of the analysis.

ELIGIBILITY:
Inclusion Criteria:

* acute self poisoning defined as the intentional intake (oral, nasal, injection etc.) of medicines during the 24h before first medical contact

Exclusion Criteria:

* cardiac arrest at first medical contact (dispatch or physician)
* acute self poisoning without any medication intake
* non intentional poisoning

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients dispatched of admitted for acute self poisoning in emergency medical services and/or emergency departments
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Percentage of each drug class | 48h

SECONDARY OUTCOMES:
odds ratio of drug classes according to sexe and age | 48h
number of participants with poisoning incident | 48h
prehospital and inhospital mortality | 30 days
percentage of each antidotal treatment | 48h
mobile intensive care unit (percentage) dispatch | 30 days
Age according to drug classes ingestion | 48h
  Median age compared according drug classes ingestion
Gender according to drug classes ingestion | 48h
  Pourcentage of gender compared according drug classes ingestion
Time (median) of admission according to drug classes ingestion | 48h
Time (median) of admission according unit of admission | 48h
Mortality according to drug class ingestion | 30 days
ICU admission according to drug class ingestion | 30 days
icu admission (percentage) | 48h
percentage of errors according to the Grenoble clinical decision rule | 30 days
multivariate analysis to describe factors associated with ICU admission | 30 days
multivariate analysis to describe factors associated with mobile intensive care unit dispatch | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Maxime Maignan, MD MSc, Principal Investigator — Emergency department, CHU Grenoble